CLINICAL TRIAL: NCT00128024
Title: Effects of Early Statin Treatment on Symptomatic Heart Failure and Ischemic Events After Acute Myocardial Infarction. The MUSASHI-AMI: A Multicenter Randomized Controlled Trial
Brief Title: Effects of Early Statin Treatment After Acute Myocardial Infarction (AMI) in Japanese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, Pofessor, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVM-RCT-2001-02; KUMSEC-2001-035
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Myocardial Infarction
Keywords: randomized prospective study; lipid-lowering therapy with any available statins; multicenter study; Japanese; acute myocardial infarction; primary percutaneous coronary intervention
MeSH Terms: conditions — Myocardial Infarction

ARMS (2):
- Statins (Active Comparator)
  Interventions: Drug: lipid-lowering treatment
- No statins (No Intervention)

INTERVENTIONS:
Drug: lipid-lowering treatment
  Arms: Statins

SUMMARY:
Statins have been shown to prevent coronary artery disease and to preserve left ventricular function in dilated cardiomyopathy. The investigators hypothesized that the early use of statins would reduce cardiovascular events including heart failure in acute myocardial infarction patients. The purpose of this study is to determine whether early (within 96 hours after onset) use of any available statins are effective to prevent cardiovascular events including heart failure after acute myocardial infarction in Japanese patients.

DETAILED DESCRIPTION:
At least, in Japanese, it was controversial if lipid-lowering therapy to the patients whose total cholesterol levels <240 mg/dL was needed. Furthermore, in general, a role for early statin therapy in patients with ST-elevated AMI reperfused by primary PCI has not been clearly established. Statins have been shown to prevent coronary artery disease and to preserve left ventricular function in dilated cardiomyopathy. The investigators hypothesized that the early use of statins would reduce cardiovascular events including heart failure in acute myocardial infarction patients. A prospective, randomized, open-label, multicenter trial is conducted in AMI patients with normal total cholesterol levels (180-240 mg/dL). Patients are randomly assigned to receive any available statin within 96 hours of AMI onset or no statin and were followed for up to 24 months. The primary endpoint is a composite of cardiovascular death, nonfatal AMI, recurrent symptomatic myocardial ischemia, congestive heart failure, and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction
* Serum total cholesterol levels on admission ranges ≥180 mg/dL and <240 mg/dL

Exclusion Criteria:

* Age < 18 years
* Time from symptom onset to admission > 96 hours
* Use of lipid-lowering agents within the previous 3 months
* Known familial dyslipidemia
* Severe renal failure
* Known hepatic disease
* Signs and symptoms of severe heart failure (Killip class III or IV)
* A scheduled PCI or coronary artery bypass grafting (CABG)
* A history of previous PCI (within 6 months) or CABG (within 3 months)
* The presence of malignant disease
* The presence of allergy to statins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2002-02; Primary Completion 2004-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
A combination of: cardiovascular death
nonfatal acute myocardial infarction
recurrent symptomatic myocardial ischemia with objective evidence and requiring emergency rehospitalization
congestive heart failure requiring emergent rehospitalization
and nonfatal stroke

SECONDARY OUTCOMES:
Reintervention procedures: coronary artery bypass grafting (CABG)
percutaneous coronary intervention (PCI) for a new lesion
and repeat PCI procedures for restenosis of the infarct-related or non-infarct-related lesions (repeat PCI occurring in the first 6 months of follow-up for an index lesion was excluded)

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, M.D., Ph.D., Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University
Locations (1):
- Department of Cardiovascular Medicine, Kumamoto University Hospital, Kumamoto, Kumamoto, Japan